CLINICAL TRIAL: NCT02662179
Title: Are the Fried Criteria Predictive of a Functional Decline in Older People With Solid Malignant Tumors?
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Murielle Surquin, Head of clinic, Brugmann University Hospital
Other Study IDs: CHUB-Fried
Record Dates: First submitted 2015-11-27; First posted 2016-01-25 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Elderly Patients With a Solid Tumor
Keywords: Elderly patients; Onco-geriatrics; Fried criteria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elderly patients with solid tumors: The group will include elderly patients with a malignant solid tumor: ovary cancer, breast cancer, digestive cancer (colo-rectal, pancreas), lung cancer or urinary tract cancer (including bladder cancer).
  Interventions: Other: Quality of life evaluation; Other: Functional decline assessment; Other: Physical decline assessment; Other: Cognitive decline assessment

INTERVENTIONS:
Other: Quality of life evaluation — Assess the quality of life ('SF-36' questionnaire) of patients 3 and 6 months after oncologic treatment. Since a diagnosis of frailness will have been established before the oncologic treatment, a correlation between the decline and the 'frail' categorization according to the Fried criteria can be established or denied.
Other: Functional decline assessment — Assess functional decline ('Katz ADL' Score and 'Lawton IADL' Score) 3 and 6 months after oncologic treatment. Since a diagnosis of frailness will have been established before the oncologic treatment, a correlation between the decline and the 'frail' categorization according to the Fried criteria can be established or denied.
Other: Physical decline assessment — Assess physical decline (walking speed and prehension force) 3 and 6 months after oncologic treatment. Since a diagnosis of frailness will have been established before the oncologic treatment, a correlation between the decline and the 'frail' categorization according to the Fried criteria can be established or denied.
Other: Cognitive decline assessment — Assess cognitive decline 3 and 6 months ('MMSE 30' questionnaire) after oncologic treatment. Since a diagnosis of frailness will have been established before the oncologic treatment, a correlation between the decline and the 'frail' categorization according to the Fried criteria can be established or denied.

SUMMARY:
Identifying the frail elderly patients or those at risk of becoming frail has become a cornerstone of modern geriatric medicine. Many instruments have been developed to identify fragility at the individual level. The 'Fragile' phenotype defined by Fried is based on 5 criteria: weakness, slowness, low level of activity, exhaustion, and unintentional weight loss. The patient is fragile if it meets at least three out of five criteria. It is 'pre-fragile' if it meets one or two criteria.

In onco-geriatrics, the International onco-geriatrics society recommends the implementation of a 'G8 scale' to detect elderly patients at risk of fragility. People with a positive G8 are then referred to the geriatric team to benefit from a comprehensive geriatric assessment. This evaluation is interpreted by the geriatrician, who proposes an action plan to overcome the various problems of the elderly patient. The evaluation can also help the oncologist in the choice of treatment for the patient: palliative care, standard treatment or adapted treatment (No-go, Go-go or slow-go).

The investigators would like to assess if fragility as defined by the Fried criteria is predictive of a functional, physical or cognitive decline, or a loss of quality of life in patients treated for a solid malignant tumor.

Furthermore, they will assess if the frailness categorization has an impact on the oncologic treatment decision. Does the oncologist switches the patient's oncologic treatment after being informed of the frailness status ?

DETAILED DESCRIPTION:
Identifying the frail elderly patients or those at risk of becoming frail has become a cornerstone of modern geriatric medicine. The term 'frail' has been elusive during quite a long time. Several studies have been conducted over the last 15 years to clarify this concept: fragility is a clinical syndrome defined by an increase of vulnerability following a decline in physiological reserves and organic functions, that compromises the ability to cope with daily life or acute stress.

Many instruments have been developed to identify fragility at the individual level. The 'Fragile' phenotype defined by Fried (Cardiovascular Health Study) is based on 5 criteria: weakness, slowness, low level of activity, exhaustion, and unintentional weight loss. The patient is fragile if it meets at least three out of five criteria. It is 'pre-fragile' if it meets one or two criteria.

In onco-geriatrics, the International onco-geriatrics society recommends the implementation of a 'G8 scale' to detect elderly patients at risk of fragility. People with a positive G8 are then referred to the geriatric team to benefit from a comprehensive geriatric assessment. This evaluation is interpreted by the geriatrician, who draws an action plan to overcome the various problems of the elderly patient. The evaluation also helps the oncologist in the choice of treatment for the patient: palliative care, standard treatment or adapted treatment (No-go, Go-go or slow-go).

However, many studies have shown that fragile patients had a greater morbidity and mortality than non-fragile patients. The rate of postoperative complications and the length of stay are significantly higher in fragile patients suffering from a colorectal cancer treated by elective surgery.

On the other hand and quite surprisingly, another study showed that none of the comprehensive geriatric assessment based fragility indicators was able to predict a post-surgery functional decline in patients having undergone surgery for colorectal cancer.

One of the primary goals of geriatry being to maintain the autonomy and independence of patients.

The investigators would thus like to assess if fragility as defined by the Fried criteria is predictive of a functional, physical or cognitive decline, or a loss of quality of life in patients treated for a solid malignant tumor.

Furthermore, they will assess if the frailness categorization has an impact on the oncologic treatment decision. Does the oncologist switches the patient's oncologic treatment after being informed of the frailness status ?

ELIGIBILITY:
Inclusion Criteria:

* Patients with a solid malign tumor: ovary cancer, breast cancer, digestive cancer (colo-rectal, pancreas), lung cancer, urinary tract cancer (including bladder cancer).
* Patients having not undergone treatment yet (be it surgery, chemotherapy or radiotherapy)
* Ambulatory or hospitalized patients

Exclusion Criteria:

* Patients unable to participate in the global geriatric evaluation (auditive or visual problems)
* Language barrier
* Clear therapeutic abstention
* Bedridden patients

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with solid tumors
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Functional decline - Katz (ADL) | 3 months after oncologic treatment
  The functional decline will be assessed by using the Katz Basic Activities of Daily Living (ADL) score
Functional decline - Katz (ADL) | 6 months after oncologic treatment
  The functional decline will be assessed by using the Katz Basic Activities of Daily Living (ADL) score
Functional decline - Lawton (IADL) | 3 months after oncologic treatment
  The functional decline will be assessed by using the Lawton Instrumental Activities of Daily Living (IADL) score
Functional decline - Lawton (IADL) | 6 months after oncologic treatment
  The functional decline will be assessed by using the Lawton Instrumental Activities of Daily Living (IADL) score
Physical decline - walking speed | 3 months after oncologic treatment
  Will be assessed by the 'Timed Up and Go' test (TUG)
Physical decline - walking speed | 6 months after oncologic treatment
  Will be assessed by the 'Timed Up and Go' test (TUG)
Physical decline - prehension force | 3 months after oncologic treatment
  Prehension force (Grip test) will be measured
Physical decline - prehension force | 6 months after oncologic treatment
  Prehension force (Grip test) will be measured
Cognitive decline - MMSE 30 | 3 months after oncologic treatment
  Will be assessed by the mini mental state evaluation (MMSE 30) questionnaire
Cognitive decline - MMSE 30 | 6 months after oncologic treatment
  Will be assessed by the mini mental state evaluation (MMSE 30) questionnaire
Quality of life - SF 36 | 3 months after oncologic treatment
  Will be assessed by the Short Form-36 (SF-36) questionnaire
Quality of life - SF36 | 6 months after oncologic treatment
  Will be assessed by the Short Form-36 (SF-36) questionnaire

SECONDARY OUTCOMES:
Switch in oncologic treatment decision | Between diagnosis and oncologic treatment - maximum 8 weeks
  Patients will be classified as frail, vulnerable or robust according to the Fried criteria. Does the oncologist changes his/her therapeutic treatment decision after being aware of the frailness categorization ?

CONTACTS AND LOCATIONS:
Overall Officials: Florence Rousseau, MD, Principal Investigator — CHU Brugmann; Murielle Surquin, MD,PhD, Principal Investigator — CHU Brugmann
Locations (2):
- Belgium (2):
  - Erasme Hospital, Brussels
  - CHU Brugmann, Brussels

REFERENCES:
- [Background] Chen X, Mao G, Leng SX. Frailty syndrome: an overview. Clin Interv Aging. 2014 Mar 19;9:433-41. doi: 10.2147/CIA.S45300. eCollection 2014. PMID 24672230
- [Background] Extermann M, Aapro M, Bernabei R, Cohen HJ, Droz JP, Lichtman S, Mor V, Monfardini S, Repetto L, Sorbye L, Topinkova E; Task Force on CGA of the International Society of Geriatric Oncology. Use of comprehensive geriatric assessment in older cancer patients: recommendations from the task force on CGA of the International Society of Geriatric Oncology (SIOG). Crit Rev Oncol Hematol. 2005 Sep;55(3):241-52. doi: 10.1016/j.critrevonc.2005.06.003. PMID 16084735
- [Background] Kristjansson SR, Nesbakken A, Jordhoy MS, Skovlund E, Audisio RA, Johannessen HO, Bakka A, Wyller TB. Comprehensive geriatric assessment can predict complications in elderly patients after elective surgery for colorectal cancer: a prospective observational cohort study. Crit Rev Oncol Hematol. 2010 Dec;76(3):208-17. doi: 10.1016/j.critrevonc.2009.11.002. Epub 2009 Dec 14. PMID 20005123
- [Background] Ronning B, Wyller TB, Jordhoy MS, Nesbakken A, Bakka A, Seljeflot I, Kristjansson SR. Frailty indicators and functional status in older patients after colorectal cancer surgery. J Geriatr Oncol. 2014 Jan;5(1):26-32. doi: 10.1016/j.jgo.2013.08.001. Epub 2013 Aug 30. PMID 24484715